CLINICAL TRIAL: NCT05115097
Title: AI Evaluation of COVID-19 Sounds
Brief Title: AI Evaluation of COVID-19 Sounds (AI-EChOS)
Acronym: AI-EChOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Emanuele Bosi, Clinical Professor, Head of Endocrino-Metabolic and Diabetologic Medicine, IRCCS San Raffaele
Other Study IDs: AI-EChOS
Record Dates: First submitted 2021-11-09; First posted 2021-11-10 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; COVID-19 Respiratory Infection; Cough; Breathing Sound; Breathing, Mouth
Keywords: COVID-19; artificial intelligence; machine learning; sound; cough; breath; voice; diagnosis; automation; AI; ML; pneumonia; symptoms; airways; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Cough; Respiratory Sounds; Mouth Breathing; Disease; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In this study the investigators record sounds of voice, breaths and cough of subjects who tested positive for COVID19. The investigators then feed these sounds into an artificial intelligence and see if it can learn to recognise features to make COVID19 diagnosis from these sounds in order to avoid to use swabs to test the general population.

ELIGIBILITY:
Inclusion Criteria:

* Adults who tested positive for SARS-CoV-2 currently admitted to hospital at the study site
* Adults who tested negative for SARS-CoV-2 and are admitted for any respiratory condition (eg COPD or asthma flare-up, pneumonia..)
* Healthy volunteers

Exclusion Criteria:

* Patients under the age of 18.
* Patients unable to read in Italian.
* Patients unable to give informed consent to participate.
* Patients requiring life support (including, but not limited to, mechanical cardiac support, ventilation, etc.)
* Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants from the general population meeting the inclusion criteria will be included in three cohorts:
  1. SARS-CoV-2 positive
  2. SARS-CoV-2 negative but with respiratory disease
  3. Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy evaluation | September 2022-December 2022
  The investigators will evaluate the accuracy of the ML algorithm in terms of sensitivity and specificity and ROC-AUC

CONTACTS AND LOCATIONS:
Overall Officials: Marco Montagna, Medicine, Principal Investigator — Vita-Salute San Raffaele University
Locations (1):
- San Raffaele Hospital and Scientific Institute, Milan, (Mi), Italy